CLINICAL TRIAL: NCT01902745
Title: Fatigue Reduction Diet in Breast Cancer Survivors
Brief Title: Fatigue Reduction Diet
Acronym: FRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Principal Investigator, Suzanna Zick, Research Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00075741
Record Dates: First submitted 2013-07-02; First posted 2013-07-18 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Chronic Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fatigue Reduction Diet (Active Comparator): The FRD maintains a participant on a diet with their typical caloric intake and replaces some of their calories with the following foods on a daily basis; whole grains, vegetables (one leafy green, one tomato, and on yellow/orange), fruit (one high in vitamin C), fatty fish and nuts and/or seeds.
  A social cognitive theory intervention method will take place that motivates the participant to change their behavior and lifestyle for overall well being.
  Interventions: Behavioral: Social Cognitive Theory
- General Health Curriculum (Active Comparator): Counseling sessions on oral health, healthy eyesight, over-the-counter drug disposal, skin and hair health, cell phone and health, hearing loss, colorectal cancer screening, and preventing colds and flu.
  A social cognitive theory intervention method will take place that motivates the participant to change their behavior and lifestyle for overall well being.
  Interventions: Behavioral: Social Cognitive Theory

INTERVENTIONS:
Behavioral: Social Cognitive Theory — Social Cognitive Theory of motivating participants to change their behaviors for overall health and well being.

SUMMARY:
There are over 2 million breast cancer survivors today. Persistent cancer-related fatigue (PCRF), a state of being tired or weary, is one of the most common and distressing symptoms experienced by breast cancer (BC) survivors. PCRF is associated with decreased quality of life, decreased sleep quality, depression, chronic pain and impaired cognition. Currently, there are few treatment options for PCRF and existing treatment options are associated with significant costs, are a considerable burden on the part of the patient, or have unacceptable side-effects. As such, there is a clear need to conduct studies evaluating the impact of safe, easy to implement and inexpensive treatments for PCRF in BC survivors.

Individualized nutritional counseling has been found to be beneficial for decreasing fatigue and improving quality of life in cancer patients receiving treatment.However, there is a dearth of research examining the use of diet for treating fatigue in cancer survivors. Our preliminary data in 40 adult cancer survivors found that fatigue severity was associated with decreased intake of key food groups, e.g., green leafy vegetables, and nutrients, e.g., omega-3 fatty acids, as reported in diet records. However, diet records are often not highly correlated with actual nutrient concentrations in the body and tend to capture short-term dietary habits not long-term patterns. The main objective of this research is to expand upon and confirm our cross-sectional preliminary data and to take advantage of a pilot clinical dietary study we are conducting by examining key nutrient differences in biological samples in the breast cancer survivors. By examining differences in biological samples we will be able to explore three key questions, which will directly influence our future interventional studies: (1) to determine if there are actual differences in concentrations of key nutrients in body tissue and which nutrients these are; (2) to assess if a dietary intervention focused on improving fatigue in BC survivors changes baseline levels of key nutrients; and (3) what is the effect size and variability of change in key nutrients in body tissue both at baseline and after a dietary intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Diagnosis of breast cancer
* Have completed all cancer related treatments (i.e. surgery, chemotherapy, radiotherapy, immunotherapy, etc.) at least 1 year prior to enrollment except hormone therapy which must have been initiated at least three weeks prior to enrollment
* Apparently cancer-free
* Have a complaint of persistent, moderate to severe fatigue despite standard treatment [defined as ≥ 4 on the Brief Fatigue Inventory (BFI)]
* Dietary eligibility requirements from a seven-day food record fruit and vegetable (FV) intake less than <5.5 servings/day, not including potatoes and iceberg lettuce.

Exclusion Criteria:

* Participants with BMI <18.5 or >35 kg/m2 will be excluded since low BMI could indicate eating disorders and high BMI values, above the midpoint of the obesity range, could indicate more prevalent health problems
* Have a diagnosis of untreated hypo- or hyper- thyroidism
* Pregnant, wanting to become pregnant or lactating women
* Unable to read and/ or write in English
* Planning on starting or stopping any chronic supplements or medications within six weeks prior to or throughout the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Fatigue in Breast Cancer Survivors | 12 weeks
  Brief Fatigue Inventory(BFI)will be filled out to assess the changes in fatigue at screening, baseline and the final 3 month visit. The BFI assesses the severity of fatigue and the impact of fatigue on daily functioning in patients with fatigue due to cancer and cancer treatment.

SECONDARY OUTCOMES:
Tolerability, Goals, Beliefs and Expectations of Participants | 12 weeks
  Tolerability, goals, beliefs and expectations of participants will be obtained through face to face conversations and over the phone. All counseling sessions will be documented into daily logs for future reference.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanna M Zick, Nd, MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Zick SM, Colacino J, Cornellier M, Khabir T, Surnow K, Djuric Z. Fatigue reduction diet in breast cancer survivors: a pilot randomized clinical trial. Breast Cancer Res Treat. 2017 Jan;161(2):299-310. doi: 10.1007/s10549-016-4070-y. Epub 2016 Dec 2. PMID 27913933